CLINICAL TRIAL: NCT05005819
Title: Evaluation of [18F]APN-1607 as a PET Biomarker for Longitudinal Change in Tau Pathology in Participants With Progressive Supranuclear Palsy
Brief Title: Evaluation of [18F]APN-1607 as a PET Biomarker
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Invicro (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APN-1607 (9646)
Record Dates: First submitted 2021-06-29; First posted 2021-08-16 (Actual); Last update posted 2025-02-20 (Actual); Status verified 2025-02

CONDITIONS: Progressive Supranuclear Palsy; Healthy Volunteers
Keywords: PSP; HV
MeSH Terms: conditions — Supranuclear Palsy, Progressive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- [18F]APN-1607 (Experimental): Participants will receive an IV bolus injection of [18F]APN-1607, followed by PET brain imaging.
  Interventions: Drug: [18F] APN-1607

INTERVENTIONS:
Drug: [18F] APN-1607 — Subjects will undergo PET imaging using [18F]APN-1607.

SUMMARY:
The overall goal of this protocol is to evaluate [18F]APN-1607 as a PET radiotracer for measuring longitudinal change in tau pathology in participants with PSP.

DETAILED DESCRIPTION:
The overall goal of this protocol is to evaluate [18F]APN-1607 as a PET radiotracer for measuring longitudinal change in tau pathology in participants with PSP. The specific objectives are:

* To characterize and demonstrate the longitudinal progression of tau deposition in vivo in participants with PSP.
* To determine optimal PET analysis parameters for [18F]APN-1607 quantification.
* To characterize the stability of tau deposition in vivo over time in healthy volunteers (HVs).
* To evaluate consistency of [18F]APN-1607 quantification in characterizing tau deposition.

ELIGIBILITY:
Inclusion Criteria for all participants:

* Males or females from 50 to 80 years of age at Screening, inclusive.
* Body weight range of ≥ 43 kg to ≤ 120 kg.
* Score ≥20 on the MMSE at Screening.
* For women of childbearing potential, agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception, and agreement to refrain from donating eggs, as defined below:

  * A woman is considered to be of childbearing potential if she is postmenarchal, has not reached a postmenopausal state (12 continuous months of amenorrhea with no identified cause other than menopause), and is not permanently infertile due to surgery (ie, removal of ovaries, fallopian tubes, and/or uterus) or another cause as determined by the Investigator (eg, Müllerian agenesis). The definition of childbearing potential may be adapted for alignment with local guidelines or regulations.
  * Women of childbearing potential must remain abstinent or use 2 methods of contraception, one of which is a barrier method (ie, male or female condom), for the study duration and 30 days after the last dose.
* Male participants with partners of childbearing potential must commit to the use of 2 methods of contraception, one of which is a barrier method (ie, male condom with or without spermicidal jelly), for the study duration and 90 days after the last dose.
* Male participants must not donate sperm for the duration of the study and 90 days after the last dose.
* For participants receiving arterial cannulation, adequate circulation to the hand for safe placement of arterial line (as determined by Allen's test) and blood clotting (prothrombin time and partial thromboplastin time [PT & PTT]).

Additional Inclusion Criteria for HVs

* Understand the study procedures and agree to participate by providing written informed consent.
* Healthy with no clinically relevant finding on physical examination at Screening.
* No cognitive impairment based on neuropsychological testing, as judged by the Investigator.
* No family history of neurological disease associated with dementia.

Additional Inclusion Criteria for Participants with PSP

* Agree to participate by providing written informed consent or written assent with informed consent from the participant's LAR or caregiver.
* Has a clinical diagnosis of probable PSP based on the National Institute of Neurological Disorders and Stroke and the Society for PSP (NINDS-SPSP) criteria (Litvan, et al 1996).
* Have Screening or prior DaTscan SPECT imaging demonstrating evidence of DaT deficit, based on visual read.
* A brain MRI scan that supports a diagnosis of PSP, with no other evidence of significant neurologic pathology.
* Deemed by the opinion of the Principal Investigator to be physically able to participate in all visits throughout the duration of the trial.
* Medications taken for symptomatic treatment of PSP should be maintained on a stable dosage regimen for at least 30 days before Screening, if possible.
* The participant has an appropriate caregiver capable of accompanying participant, if applicable.

Exclusion Criteria for all participants:

* Participants are only eligible if they do not fulfill any of the exclusion criteria for the participant group.

  * Current or prior history (in the last 12 months) of any alcohol or drug abuse.
  * Laboratory tests with clinically significant abnormalities and/or clinically significant unstable medical illness.
  * Participants with QT interval corrected for heart rate using Fridericia's formula (QTcF) >450 msec (males) or >470 msec (females) at Screening will be excluded. ECG measurements may be repeated once.
  * Has received an investigational drug or device within 30 days of Screening.
  * Prior participation in other research protocols or clinical care in the last year in addition to the radiation exposure expected from participation in this clinical study, such that radiation exposure exceeds the effective dose of 50 mSv, which would be above the acceptable annual limit established by the US Federal Guidelines.
  * Pregnancy, lactating or breastfeeding.
  * Evidence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, neoplastic, endocrine, alternative neurological, immunodeficiency, pulmonary, or other disorder or disease.
  * Unsuitable veins for repeated venipuncture or contraindication to arterial blood sampling (for participants who will receive arterial blood sampling).
  * MRI exclusion criteria include: Findings that may be responsible for the neurologic status of the participant such as significant evidence of cerebrovascular disease (more than 2 lacunar infarcts, any territorial infarct >1 cm3, or deep white matter abnormality corresponding to an overall Fazekas scale of 3 with at least one confluent hyperintense lesion on the fluid-attenuated inversion recovery (FLAIR) sequence that is ≥20 mm in any dimension), infectious disease, space-occupying lesions, normal pressure hydrocephalus or any other abnormalities associated with central nervous system (CNS) disease (other than findings consistent with PSP for participants with PSP).
  * Implants such as implanted cardiac pacemakers or defibrillators, insulin pumps, cochlear implants, metallic ocular foreign body, implanted neural stimulators, CNS aneurysm clips and other medical implants that have not been certified for MRI, or history of claustrophobia in MRI.
  * Use of over the counter (OTC) medication (except acetaminophen), dietary supplements, or vitamins, within 2 weeks prior to initial dosing, unless approved by the Investigator.
  * Has a known hypersensitivity to any component of the formulation of [18F]APN-1607 or related compounds.
  * Major surgery, or donation or loss of 400 mL or more of blood within 4 weeks prior to initial dosing, or longer, if required by local regulation.
  * History of immunodeficiency diseases, including a positive HIV test result.
  * A positive Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody test result.
  * Participant is, in the opinion of the Investigator, unsuitable in any other way to participate in this study.
  * If available, evidence of amyloid deposition on amyloid PET.
  * Any new or change in prescription drugs prior to initial dosing, unless approved by the Investigator.

Additional Exclusion Criteria for HVs

• The participant is currently exposed to nicotine products or had regular nicotine exposure within a six-month period, to be verified by urine cotinine screening

Additional Exclusion Criteria for Participants With PSP

* Ongoing treatment with methylphenidate, modafinil, metoclopramide, alpha methyldopa, reserpine, or amphetamine derivative, for participants requiring DaTscan imaging.
* Participant has known hypersensitivity to iodine or potassium iodide (KI) in the opinion of the Investigator.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2024-01-09 (Actual); Study Completion 2024-01-09 (Actual)

PRIMARY OUTCOMES:
Change in standardized uptake value ratios (SUVRs) of regional [18F]APN-1607. | 72 weeks
  The within-group change in standardized uptake value ratios (SUVRs) of regional [18F]APN-1607 binding within a priori defined cortical and subcortical brain regions from Baseline to Week 36 and Week 72.

CONTACTS AND LOCATIONS:
Overall Officials: David Russell, M.D., Ph.D., Principal Investigator — Invicro
Locations (1):
- Invicro, New Haven, Connecticut, United States

REFERENCES:
- See also: Related Information — http://invicro.com